CLINICAL TRIAL: NCT02352402
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Investigating The Effect Of Ticagrelor On Saphenous Vein Graft Patency In Patients Undergoing Coronary Artery Bypass Grafting Surgery (The POPular CABG Study)
Brief Title: The Effect Of Ticagrelor On Saphenous Vein Graft Patency In Patients Undergoing Coronary Artery Bypass Grafting Surgery
Acronym: POPular CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: J.M. ten Berg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, J.M. ten Berg, MD, PhD, FESC, FACC, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POPCABG; 2014-002142-50 (EudraCT Number)
Record Dates: First submitted 2014-09-19; First posted 2015-02-02 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease; Stable Angina; Acute Coronary Syndrome
Keywords: CABG; Ticagrelor; Graft; Patency
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90mg twice daily for 1 year on top of ASA
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator): Placebo matching ticagrelor 90mg twice daily on top of ASA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor
  Other Names: Brilique; Brillinta
  Arms: Ticagrelor
Drug: Placebo
  Arms: Placebo

SUMMARY:
In the POPular CABG study we investigate if the addition of ticagrelor, a drug that inhibits blood platelets from clotting, to treatment with aspirin will reduce the rate of saphenous vein graft occlusion as assessed with coronary computed tomography angiography at 1 year after coronary artery bypass grafting surgery.

DETAILED DESCRIPTION:
Rationale: Acetylsalicylic acid (ASA) is used to prevent the occlusion of grafts placed during coronary artery bypass grafting surgery (CABG) and to reduce the incidence of atherothrombotic events during follow-up. Graft occlusion occurs predominantly in saphenous vein grafts (SVGs) and can result in symptoms of chest pain, myocardial infarction (MI) and even death. The anti-thrombotic effect of ASA is a result of the inhibition of the generation of thromboxane A2 (TXA2) in blood platelets. Despite ASA therapy, 6.8% to 26% of SVGs occlude in the first year after CABG, mainly due to thrombus formation. This might be due to the fact that ASA is not equally effective in all patients, indicated by a substantial amount of patients that still generate TXA2 and show activated platelets, despite adequate ASA use. We hypothesize that more potent platelet inhibition by the addition of ticagrelor to standard ASA therapy could decrease the rate of SVG occlusion.

Main objective: To investigate whether a combination of ticagrelor 90mg twice daily and ASA 80mg once daily is superior to ASA 80mg once daily alone in the prevention of SVG occlusion in patients who underwent CABG with use of one or more SVGs, as assessed with coronary computed tomography angiography (CCTA) at 1 year after randomization.

Study design: Randomized, double-blind, placebo-controlled, multicenter trial. Number of patients: Approximately 500 patients will be randomized.

Study population: Patients undergoing CABG with one or more SVGs, CABG being an isolated procedure or part of combined surgery.

Informed consent procedure, screening and sample size: We will screen patients and obtain informed consent before CABG. After CABG patients who gave informed consent are screened again to check if the patient fulfills the inclusion criteria and does not have any exclusion criteria. A total of 500 patients will receive randomized study medication after CABG.

Intervention: Patients will be randomly assigned to treatment with 90mg of ticagrelor or a matching placebo twice daily in addition to standard treatment with ASA for the duration of 1 year. Patients will be prescribed 80mg of ASA once daily according to routine clinical practice. Graft patency will be assessed with CCTA 1 year after randomization. If the patient consents to participate in the substudies, platelet function tests will be performed before surgery and 3 days and 1 year after randomization. Thirty day and one-year follow-up of clinical events will be obtained for all patients by screening the (electronic) patient file, telephonic interviews, study site visits and possibly with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* More than 21 years of age
* Planned coronary artery bypass grafting (CABG) with the use of 1 or more saphenous vein grafts, CABG being an isolated procedure or part of a combined aortic valce replacement surgery with bioprothesis.

Exclusion Criteria:

* Unable to give informed consent or a life expectancy of less than 1 year
* Concomitant valve, aorta or rhythm surgery during the same session, (excluding aortic bioprothesis)
* Inability to undergo coronary computed tomography angiography, in the investigator's opinion, for instance due to severe claustrophobia or contrast allergy
* Use of oral anticoagulants (acenocoumarol, phenprocoumon, dabigatran, rivaroxaban, etc) and a contraindication for discontinuation of this medication or the expectation that the patient will have an indication for the use of these drugs after surgery
* Placement of a drug-eluting stent in a coronary or cerebral artery within 6 months of CABG or placement of a bare-metal stent in a coronary or cerebral artery within 1 month of CABG
* Use of antiplatelet drugs other than aspirin (clopidogrel, prasugrel, ticagrelor, dipyridamol, etc.) and a contraindication for discontinuation of this medication after CABG, according to the treating physician or the investigator
* Women who are known to be pregnant, who have given birth within the past 90 days or who are breastfeeding
* Pre-menopausal women without adequate contraception
* Severe renal function impairment requiring dialysis
* Moderate or severe hepatic impairment
* Active malignancy with increase in bleeding risk, in the investigator's opinion
* Use of strong inhibitors of CYP3A4 (e.g. ketaconazole, clarithromycin, nefazodone, ritonavir, atazanavir)
* Clinically significant out of range values for platelet count or haemoglobin at screening, in the investigator's opinion
* Contraindication for the use of ticagrelor or aspirin (i.e. history of intracranial bleeding, high bleeding risk, previous allergic reaction), in the investigator's opinion
* Previous inclusion in this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Saphenous vein graft occlusion | 1 year after coronary artery bypass grafting
  As assessed with coronary computed tomography angiography or clinically indicated coronary angiography

SECONDARY OUTCOMES:
Saphenous vein graft failure | 1 year after coronary artery bypass grafting
  Composite of saphenous vein graft occlusion as assessed with coronary computed tomography angiography or clinically indicated coronary angiography, saphenous vein graft revascularization, myocardial infarction in the myocardial territory supplied by a saphenous vein graft or sudden death
Significant saphenous vein graft stenosis | 1 year after coronary artery bypass grafting
  As assessed with coronary computed tomography angiography or clinically indicated coronary angiography
BARC minor (type 1 or 2) and major (type 3, 4 or 5) bleeding | 30 days after coronary artery bypass grafting
  Bleeding Academic Research Consortium bleeding criteria
BARC minor (type 1 or 2) and major (type 3, 4 or 5) bleeding | 1 year after coronary artery bypass grafting
  Bleeding Academic Research Consortium bleeding criteria
TIMI minor and major bleeding | 30 days after coronary artery bypass grafting
  Thrombolysis in Myocardial Infarction bleeding criteria
TIMI minor and major bleeding | 1 year after coronary artery bypass grafting
  Thrombolysis in Myocardial Infarction bleeding criteria
High platelet reactivity | Within 72h before coronary artery bypass grafting
  As assessed with platelet function tests.
High platelet reactivity | 3 days after coronary artery bypass grafting
  As assessed with platelet function tests.
High platelet reactivity | 1 year after coronary artery bypass grafting
  As assessed with platelet function tests.
Level of GDF-15 | Within 72h before coronary artery bypass grafting
  Growth differentiation factor 15 level
Level of GDF-15 | 3 days after coronary artery bypass grafting
  Growth differentiation factor 15 level
Level of GDF-15 | 1 year after coronary artery bypass grafting
  Growth differentiation factor 15 level
Arterial graft occlusion | 1 year after coronary artery bypass grafting
  As assessed with coronary computed tomography angiography or clinically indicated coronary angiography
All graft occlusion | 1 year after coronary artery bypass grafting
  As assessed with coronary computed tomography angiography or clinically indicated coronary angiography
Significant arterial graft stenosis | 1 year after coronary artery bypass grafting
  As assessed with coronary computed tomography angiography or clinically indicated coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën M ten Berg, MD, PhD, Study Chair — St. Antonius Hospital
Locations (6):
- Netherlands (6):
  - St Antonius Hospital, Nieuwegein, Utrecht
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud UMC, Nijmegen
  - Erasmus Erasmus UMC, Rotterdam

REFERENCES:
- [Background] Willemsen LM, Janssen PWA, Hackeng CM, Kelder JC, Tijssen JGP, van Straten AHM, Soliman-Hamad MA, Deneer VHM, Daeter EJ, Sonker U, Klein P, Ten Berg JM. A randomized, double-blind, placebo-controlled trial investigating the effect of ticagrelor on saphenous vein graft patency in patients undergoing coronary artery bypass grafting surgery-Rationale and design of the POPular CABG trial. Am Heart J. 2020 Feb;220:237-245. doi: 10.1016/j.ahj.2019.12.001. Epub 2019 Dec 13. PMID 31884246
- [Derived] Willemsen LM, Janssen PWA, Peper J, Soliman-Hamad MA, van Straten AHM, Klein P, Hackeng CM, Sonker U, Bekker MWA, von Birgelen C, Brouwer MA, van der Harst P, Vlot EA, Deneer VHM, Chan Pin Yin DRPP, Gimbel ME, Beukema KF, Daeter EJ, Kelder JC, Tijssen JGP, Rensing BJWM, van Es HW, Swaans MJ, Ten Berg JM. Effect of Adding Ticagrelor to Standard Aspirin on Saphenous Vein Graft Patency in Patients Undergoing Coronary Artery Bypass Grafting (POPular CABG): A Randomized, Double-Blind, Placebo-Controlled Trial. Circulation. 2020 Nov 10;142(19):1799-1807. doi: 10.1161/CIRCULATIONAHA.120.050749. Epub 2020 Aug 31. PMID 32862716
- [Derived] Feitosa MPM, Soffiatti CD, Linhares Filho JPP, Batista DV, Lobo Filho HG, Lima EG, Serrano Junior CV. Dual platelet antiaggregation therapy after myocardial revascularization surgery. Rev Assoc Med Bras (1992). 2019 Mar;65(3):316-318. doi: 10.1590/1806-9282.65.3.316. Epub 2019 Apr 11. PMID 30994825